CLINICAL TRIAL: NCT03730584
Title: Evaluation of the Efficacy of a Topical Analgesic Treatment With ROPIVACAINE in Children and Young Adults With Hereditary Epidermolysis Bullosa
Brief Title: Evaluation of the Efficacy of ROPIVACAINE in Children and Young Adults With Hereditary Epidermolysis Bullosa
Acronym: EBROPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20180207; 2018-003334-33 (EudraCT Number)
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Epidermolysis Bullosa
Keywords: Hereditary Epidermolysis Bullosa; pain; bath; dressing change; Ropivacaine; topical application
MeSH Terms: conditions — Epidermolysis Bullosa; Pain | interventions — Ropivacaine; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Hereditary Epidermolysis Bullosa (Experimental)
  Interventions: Drug: Ropivacaine; Biological: Blood test

INTERVENTIONS:
Drug: Ropivacaine — Ampoules of ROPIVACAINE 2mg / ml will be used by local cutaneous application in soft application with device of "hand shower" on the painful wounds without exceeding the dose of 1mg / kg per bath.
Biological: Blood test — Blood test during the first bath with Ropivacaine for Titration of Ropivacaine

SUMMARY:
The purpose of this study is to determine whether topical application of Ropivacaine is effective for treating refractory pain during dressing changes and so improve quality of life of patients (newborn, child, adolescent or adults under 21) suffering from hereditary epidermal epidermolysis bullosa.

DETAILED DESCRIPTION:
This clinical trial aims to determine the efficacy on pain of local application of ROPIVACAINE 0.2% on cutaneous lesions related to Epidermolysis Bullosa during dressing change, associated with the standard premedication.

Patients will be hospitalized and will have several baths. The first bath will be done according to usual protocol (usual premedication 1h before the bath). Pain measurements (Visual analog scale or FLACC) will be done at the entry into the water, in the middle of bath and at the time of the dressing change.

The following baths will be done using local application of Ropivacaine 15 minutes before entering into the water on lesions identified by the patients as the most painful lesions due to Epidermolysis Bullosa.

A blood test will be done during the first use of Ropivacaine to determine plasmatic level of Ropivacaine.

After 3 baths in the dermatology unit, patients will continue such bath at home, every 48h during 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Minor patient or adult ≤ 21 years of age with hereditary epidermolysis bullosa,
* Presenting pain at the entrance of the bath with an average of EVA or FLACC greater than 4/10 the week before the inclusion
* Usually requiring premedication with weak or strong opioid
* Parental consent if minor or patient consent
* Affiliated with Social Security

Exclusion Criteria:

* Patient with a known allergy to ROPIVACAINE or other local anesthetics with amide binding or one of the excipients mentioned in the SPC
* Severe renal insufficiency defined by DFG below 29ml / min
* Moderate to severe hepatic insufficiency defined by a Child-Pugh B or C score and AST or ALAT greater than 3 times normal
* Moderate to severe cardiac failure defined by FEGV less than 45% and/or NYHA class II to IV
* Hypovolemia

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Efficacy on pain of Ropivacaine at the bath entrance | Day 5
  Evaluation performed by child with a Visual Analog Scale (VAS) or by parents with the Face Legs Activity Cry Consolability questionary (FLACC) - defined by a 2 points loss between day 1 and day 5

SECONDARY OUTCOMES:
Efficacy on pain of Ropivacaine at the time of dressing change | Day 5
  Evaluation performed by child with a VAS or by parents with FLACC at the time of dressing changes after bathing - defined by a 2 points loss between day 1 and day 5
Efficacy on pain of Ropivacaine at home at the time of dressing change | Day 21
  Evaluation performed by child with a VAS or by parents with FLACC at the time of dressing changes after bathing
Efficacy on pain of Ropivacaine at home at bath entrance | Day 21
  Evaluation performed by child with a VAS or by parents with FLACC at the time of bath entrance
Measurement of Local or systemic side effects | Day 5
  Evaluation of tolerance of Ropivacaine
Efficacy of Ropivacaine on the reduction of opioids use | Day 21
  Efficacy of ROPIVACAINE on the reduction of weak or strong opioids consumption for premedication for the bath and dressing change
Efficacy of Ropivacaine on the reduction of benzodiazepines or hypnotics use | Day 21
  Efficacy of ROPIVACAINE on the reduction of of benzodiazepines or hypnotics consumption for premedication for the bath and dressing change
Systemic passage of Ropivacaine | Blood test during the first bath with Ropivacaine up to Day 4
  Evaluation of the systemic passage of Ropivacaine

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bodemer, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Céline Greco, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moreno Artero E, Schinkel N, Chaumon S, Corset I, Rabeony T, Elie C, Bellon N, Bodemer C, Greco C. Efficacy of topical ropivacaine in children and young adults with hereditary epidermolysis bullosa. Br J Dermatol. 2021 Mar;184(3):550-552. doi: 10.1111/bjd.19551. Epub 2020 Nov 2. No abstract available. PMID 32939751
- [Result] Chevret S, Verlhac S, Ducros-Miralles E, Dalle JH, de Latour RP, de Montalembert M, Benkerrou M, Pondarre C, Thuret I, Guitton C, Lesprit E, Etienne-Julan M, Elana G, Vannier JP, Lutz P, Neven B, Galambrun C, Paillard C, Runel C, Jubert C, Arnaud C, Kamdem A, Brousse V, Missud F, Petras M, Doumdo-Divialle L, Berger C, Freard F, Taieb O, Drain E, Elmaleh M, Vasile M, Khelif Y, Bernaudin M, Chadebech P, Pirenne F, Socie G, Bernaudin F. Design of the DREPAGREFFE trial: A prospective controlled multicenter study evaluating the benefit of genoidentical hematopoietic stem cell transplantation over chronic transfusion in sickle cell anemia children detected to be at risk of stroke by transcranial Doppler (NCT 01340404). Contemp Clin Trials. 2017 Nov;62:91-104. doi: 10.1016/j.cct.2017.08.008. Epub 2017 Aug 15. PMID 28821470